CLINICAL TRIAL: NCT02369536
Title: Clinical Trial on the Efficacy of a Natural Components Mixture in the Treatment of Non Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Efficacy of a Natural Components Mixture in the Treatment of Non Alcoholic Fatty Liver Disease (NAFLD)
Acronym: NUTRAFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Giovanni de Gaetano, Head, Department Epidemiology and Prevention, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neuromed-Nutrafast-PON2015
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: NAFLD; nutraceutical mixture
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nutraceutical mixture (Active Comparator): Lifestyle counseling plus three month administration of nutraceutical mixture (2 soft gelatin capsules of 800 mg per day)
  Interventions: Dietary Supplement: nutraceutical mixture
- placebo (Placebo Comparator): Lifestyle counseling plus three month administration of placebo formulation (2 soft gelatin capsules of 800 mg per day)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: nutraceutical mixture — Lifestyle counseling, administration of a nutraceutical mixture: fish oil 70% DHA (docosahexaenoic acid), phosphatidylcholine concentrated in sunflower oil, silymarin, choline bitartrate, curcumin, D-α-tocopherol; choline (82,5 mg, corresponding to 15% of the average intake of 550 mg per day in an adult man)
  Arms: nutraceutical mixture
Dietary Supplement: placebo — Lifestyle counseling, administration of a placebo, containing only choline, at the same low concentration of the active mixture
  Arms: placebo

SUMMARY:
The objective of this study is to provide clinical data to support the effectiveness of a mixture of ingredients of natural origin, suitably selected and packaged, in the protection from liver damage, in subjects with NAFLD.

Study design: double-blind, randomized, multicentre trial, placebo-controlled on two parallel groups.

The study participants are healthy volunteers, since they do not have nor had any liver-related clinical symptom, but simply laboratory (plasma levels greater than normal for at least one of the liver parameters -aspartate aminotransferase AST, alanine aminotransferase ALT or γ -glutamyltranspeptidase γ-GT) or instrumental (ultrasonographic abnormalities of steatosic liver) tests altered as compared to normal ranges.

Three months treatment with the nutraceutical mixture or placebo. Outcomes tested before and at the end of treatment - 3 months).

DETAILED DESCRIPTION:
A correct hepatic function is highly relevant from the epidemiological point of view. In Italy, Non Alcoholic Fatty Liver Disease - NAFLD - has a prevalence of 20-25% in the adult population, with peaks of 50-70% within obese and type-2 diabetes populations: it is the most frequent cause of hematic changes in cytonecrosis enzymes, and can explain about 90% of asymptomatic high levels of transaminases. NAFLD natural history is associated with an increase of cerebro and cardiovascular risk, in both healthy subjects and diabetic patients.

Its prevention and treatment are of great interest, in particular dietary and nutraceutical interventions are the object of innovative research. It is also known that about 65% of subjects with hepatic dysfunction consume plant extracts, like silymarin from Cardo marianum. A recent trial showed an improvement of the hepatic function in subjects with NAFLD treated with silybin, combined with phosphatidylcholine and vitamin E. These findings provide valuable information on new therapeutic strategies, but warrant further investigation. For no natural substance a health claim related to liver function was in fact approved by the European Food Safety Authority (EFSA). The only exception is constituted by the food sources of choline, for which the maintenance of normal hepatic function has been claimed.

The objective of this study is to provide clinical data to support the effectiveness of a mixture of ingredients of natural origin, suitably selected and packaged, in the protection from liver damage, in subjects with NAFLD.

Treatment: subjects will be randomized to receive the nutraceutical formulation or placebo for three months, in the amount of two capsules (about 800 mg each) a day, at one time.

All subjects, after signing a written informed consent to participation in the study, will receive appropriate recomendations about diet and physical exercise.

A clinic visit, with collection of the patient clinical and pharmacological history and recording of any adverse event, liver ultrasound, measurement of weight and height and calculation of BMI, measure of arterial blood pressure, collection of a sample of venous blood, under fasting conditions, for hematochemical tests, will be made at the baseline (T0); all examinations and tests (except liver ultrasound) will be repeated after three months of treatment (T1).

Primary end-points of the study: hematic levels of hepatic enzymes: ALT, AST and γ-GT.

Secondary end-points of the study:

1. Hepatic function: direct and indirect bilirubin;
2. Inflammation markers: C Reactive Protein (CRP), interleukin (IL)-6, IL-1β, IL-8, IL-10, Receptor for Advanced Glycation End Products (RAGE), Advanced Glycation End Products (AGE), insulin-like growth factor-1 (IGF-1)
3. Haemostatic function: Factor VII, fibrinogen, thrombin generation with and without thrombomodulin, antithrombin (AT), tissue-type Plasminogen Activator (t-PA), Plasminogen Activator Inhibitor-1(PAI-1), thrombin activatable fibrinolysis inhibitor (TAFI) and activated TAFI (TAFIa), plasmin-antiplasmin complex, plasma fibrinolytic capacity;
4. Metabolic syndrome parameters: glycemia, triglycerides, HDL cholesterol, insulin e insulin-resistance (HOMA-IR homeostasis model assessment-estimated insulin resistance), adiponectin;
5. Apoptosis parameters: total cytokeratin-18 (M65 antigene), M30 and M65/M65ED, soluble fas and soluble fas ligand.

A weekly food diary will be administered to each subject before and at the end of the treatment, to highlight any possible change of dietary habits during the study.

In addition, for all subjects the NAFLD Fibrosis Score (NFS), a composite score of prognostic value for the conversion of NAFDL into fibrotic hepatitis and for the disease severity, will be calculated. This score includes age, body mass index, platelet count, albumin, relationship between AST and ALT, and presence of diabetes. A sub-analysis will be done to evaluate the efficacy of the treatment with the synergistic blend of ingredients in subjects with high, as compared to those with low NFS.

Sample size calculation: Establishing Alpha = 0.05 and Β = 80%, the number of 150 people (75 per treatment arm) will evaluate differences between the two groups (T1 to T0) equal to 46% of the standard deviation of the mean of the two liver function parameters selected (primary end-points), in particular, differences over 11.5 for ALT (17% of the average), 7.1 for AST (17% of the average) or 13.8 for γ-GT (19% of the average). This calculation also includes a drop-out of 10% of the sample enrolled in the study.

Compliance to treatment will be monitored by counting the capsules returned in the box at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* subjects with non alcoholic fatty liver disease (NAFLD)
* presenting ultrasonographic abnormalities of steatosic liver (hyperechogenic parenchyma)
* with plasma levels greater than normal (ranges of each recruiting center) for at least one of the following parameters (aspartate aminotransferase AST, alanine aminotransferase ALT, γ -glutamyltranspeptidase γ-GT).

Exclusion Criteria:

* history of alcohol abuse
* use of drugs associated with the development of hepatic steatosis
* malnutrition
* alcoholic chronic liver disease
* chronic liver disease of different etiology (autoimmune disease, primary biliary cirrhosis, primary sclerosing cholangitis, hereditary hemochromatosis, Wilson's disease, deficits of alpha-1 antitrypsin, celiac disease)
* severe renal, cardiac or respiratory insufficiency
* malignant tumors
* intolerance to any component of the active ingredients of the formulation
* women who are pregnant or have planned the pregnancy within three months and women who are breast-feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni de Gaetano, MD PhD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ; American Association for the Study of Liver Diseases; American College of Gastroenterology; American Gastroenterological Association. The diagnosis and management of non-alcoholic fatty liver disease: Practice guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Am J Gastroenterol. 2012 Jun;107(6):811-26. doi: 10.1038/ajg.2012.128. No abstract available. PMID 22641309

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nutraceutical Mixture | Placebo
Started | 62 | 64
Completed | 55 | 58
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutraceutical Mixture | Placebo | Total
Number analyzed (Participants) | 55 | 58 | 113
Age, Categorical [Count of Participants; unit: Participants] — Population: Subjects lost at follow-up: 7 in the active group and 6 in the control group.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 47 | 47 | 94
    >=65 years | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Subjects lost at follow-up:
  7 in the active group, for: bone fracture (1), relocation to another city (1), discontinued supplementation for dermatitis (1), unmotivated personal decision (4);
  6 in the control group, for: discontinued supplementation for faecal color abnormality (green faeces, 1), unmotivated personal decision (5)
  years | 55.7 (12.2) | 53.4 (11.3) | 54.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Subjects lost at follow-up: 7 in the active group and 6 in the control group.
  Participants
    Female | 20 | 19 | 39
    Male | 35 | 39 | 74
Region of Enrollment [Number; unit: participants] — Population: Subjects lost at follow-up: 7 in the active group and 6 in the control group.
  participants
    Italy | 55 | 58 | 113

OUTCOME MEASURES:

1. Primary Outcome: Hematic Levels of Hepatic Enzymes AST
Description: hematic levels of hepatic enzyme: aspartate aminotransferase (AST)
Time Frame: before and at the end of treatment (three months)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Nutraceutical Mixture | Placebo
Number analyzed (Participants) | 55 | 58
IU/L
  before treatment | 35.4 (22.5) | 37.5 (25.2)
  after 3 months | 31.6 (15) | 31.2 (14.7)
Statistical Analysis 1: Comparison: Nutraceutical Mixture vs Placebo; Intention-to-treat-analysis. Differences between basal values in active and control groups and between T1 vsT0 changes in the two groups assessed by ANOVA and Fisher's exact test; Test type: Superiority or Other; p < 0.05, ANOVA

2. Primary Outcome: Hematic Levels of Hepatic Enzymes ALT
Description: hematic levels of hepatic enzyme: alanine aminotransferase (ALT)
Time Frame: before and at the end of treatment (three months)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Nutraceutical Mixture | Placebo
Number analyzed (Participants) | 55 | 58
IU/L
  before treatment | 45.5 (28.4) | 48.3 (43.4)
  after 3 months | 43.8 (22.9) | 40.0 (21.9)

3. Primary Outcome: Hematic Levels of Hepatic Enzymes GGT
Description: hematic levels of hepatic enzyme: gamma-glutamyl transpeptidase (GGT)
Time Frame: before and at the end of treatment (three months)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Nutraceutical Mixture | Placebo
Number analyzed (Participants) | 55 | 58
IU/L
  before treatment | 101.4 (101.0) | 98.5 (136.0)
  after 3 months | 87.2 (71.1) | 75.6 (64.4)

4. Secondary Outcome: Plasma Levels of Hepatic Enzymes
Description: hematic levels of direct bilirubin
Time Frame: before and at the end of treatment (three months)
Population: direct bilirubin
Measure: Mean (Standard Deviation); unit: microM/L
Arm/Group | Nutraceutical Mixture | Placebo
Number analyzed (Participants) | 55 | 58
microM/L
  before treatment | 2.05 (1.2) | 2.74 (2.91)
  3 months after | 2.22 (1.2) | 2.39 (1.71)
Statistical Analysis 1: Comparison: Nutraceutical Mixture vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, ANOVA

5. Secondary Outcome: Levels of Circulating Inflammation Marker
Description: Levels of circulating Inflammation marker: C Reactive Protein (CRP)
Time Frame: before and at the end of treatment (three months)
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Nutraceutical Mixture | Placebo
Number analyzed (Participants) | 55 | 58
nmol/L
  before treatment | 21.0 [13.3 to 38.1] | 28.3 [3.4 to 44.5]
  3 months after | 17.1 [12.9 to 30.5] | 24.0 [13.3 to 41.0]

6. Secondary Outcome: Measures of the Haemostatic Function
Description: Tissue-type Plasminogen Activator (t-PA) levels in plasma
Time Frame: before and at the end of treatment (three months)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Nutraceutical Mixture | Placebo
Number analyzed (Participants) | 55 | 58
ng/ml
  before treatment | 8.6 (4.8) | 10.1 (9.0)
  after 3 months | 8.7 (4.9) | 9.9 (8.9)

7. Secondary Outcome: Measures of the Haemostatic Function
Description: Plasminogen Activator Inihibitor (PAI-1) levels in plasma
Time Frame: before and at the end of treatment (three months)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Nutraceutical Mixture | Placebo
Number analyzed (Participants) | 55 | 58
ng/ml
  before treatment | 42.7 (19.8) | 48.0 (18.5)
  after 3 months | 44.3 (18.4) | 47.7 (21.9)

8. Secondary Outcome: Measures of the Haemostatic Function
Description: Thrombin activatable fibrinolysis inhibitor (TAFI) levels in plasma
Time Frame: before and at the end of treatment (three months)
Measure: Mean (Standard Deviation); unit: % of reference plasma
Arm/Group | Nutraceutical Mixture | Placebo
Number analyzed (Participants) | 55 | 58
% of reference plasma
  before treatment | 105 (23) | 100 (23)
  after 3 months | 104 (23) | 99 (21)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Nutraceutical Mixture | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/58
Other Adverse Events (participants affected / at risk) | 0/55 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No